CLINICAL TRIAL: NCT00492843
Title: A Randomized Study to Evaluate the Safety and Efficacy of Loading Dose of Bondronat Versus Standard Dose of Bondronat in Patients With Lung Cancer and Skeletal Metastasis Experiencing Moderate to Severe Pain
Brief Title: Loading Dose or Standard Dose of Intravenous Ibandronate in Treating Patients With Lung Cancer and Skeletal Metastasis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It is too difficult to recruit suitable patients.
Sponsor: Chinese Society of Lung Cancer (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Professor, Chinese Society of Lung Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSLC0701
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer
Keywords: Ibandronate, Lung cancer, bone metastasis
MeSH Terms: conditions — Lung Neoplasms | interventions — Ibandronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Intravenous infusion of either 6mg Bondronat on three consecutive days
  Interventions: Drug: Ibandronate (Bondronat)
- B (Active Comparator): Intravenous infusion of 6mg Bondronat on one day
  Interventions: Drug: Ibandronate (Bondronat)

INTERVENTIONS:
Drug: Ibandronate (Bondronat) — Intravenous infusion of either 6mg Bondronat on three consecutive days or 6mg Bondronat on one day.
  Other Names: no other names

SUMMARY:
The objective of this trial is to assess the efficacy and safety of loading doses versus standard dose of intravenous Bondronat in reducing pain in patients with lung cancer and bone metastatic disease.

DETAILED DESCRIPTION:
Patients with lung cancer and bone metastatic disease may experience moderate or severe bone pain. Some researches have reported that loading doses Bondronat (6mg Bondronat on three consecutive days) had great efficacy in reducing pain in patients with malignant bone disease without unacceptable toxicities. So,we designed this clinical trial to compare the efficacy and safety profiles between loading doses Bondronat and standard dose Bondronat.Enrolled patients will receive an intravenous infusion of either 6mg Bondronat on three consecutive days or 6mg Bondronat on one day. The targeted sample size is 120 individuals. Primary outcome measures will be bone pain response ( ≥ 25% decrease in mean pain score with a maximum of 15% increase in mean analgesic consumption). Secondary outcome measures will be efficacy including ECOG Performance status, analgesic consumption, bone markers, and safety profiles including AE and laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Histological or cytological evidence of lung cancer
* Presence of bone metastases documented on bone X-ray, bone ECT, CT scan or MRI scan
* Mean pain score ≥ 4 during 3-day baseline period on the WORSE pain scale of the VAS
* Patients must be on a stable dose of analgesics over the 3-day baseline period (maximum 15% variation is allowed)
* ECOG Performance status of 0-3 (patients with PS of 3 must have their score based on bone pain, not underlying neoplastic disease)
* Adequate renal function: creatinine clearance ≥ 50 ml/min (cockroft formula) and serum creatinine ≤ 2.0mg/dl (168 µmol/L); ALT or AST within 2 times the upper limit of the normal range

Exclusion Criteria:

* Patients with an uncontrolled infection
* Hypocalcemia
* Patients who have received a bisphosphonate within 3 weeks of the start of the Baseline period or who are currently receiving another bisphosphonate
* Patients with known hypersensitivity to any of the components of ibandronic acid
* Patients who are pregnant or lactating
* Radiotherapy to bone within the 28 days prior inclusion or during the trial duration
* Patient who are currently treated with any other investigational therapy or have received it within 30 days of the first schedule day of dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
bone pain response (≥25% decrease in mean pain score with a maximum of 15% increase in mean analgesic consumption) | 1 month

SECONDARY OUTCOMES:
Efficacy: ECOG Performance status, Analgesic consumption, bone marker Safety: AE, laboratory parameters | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (8):
- China (8):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The Tumor Hospital of Harbin Medical University, Harbin
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - General Hospital of Tianjin Medical University, Tianjin

REFERENCES:
- See also: Related Info — http://www.lungca.com